CLINICAL TRIAL: NCT05345470
Title: Dose Response Effect of Chia Seeds on Subjective Appetite and Glycemic Response: a Single Center, Randomized Cross-over Study in Healthy Adults
Brief Title: Dose Response Effect of Chia Seeds on Subjective Appetite and Glycemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2117
Record Dates: First submitted 2022-04-18; First posted 2022-04-26 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Nutrition, Healthy
Keywords: chia seeds; chia; Salvia hispanica L.; hunger; fullness; satiety; glycemic response

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0 grams of chia seeds (Placebo Comparator): 3 cookies (30 grams)
  Interventions: Other: 140 calories per 30 gram test meal
- 3 grams of chia seeds (Experimental): 3 cookies (30 grams)
  Interventions: Other: 140 calories per 30 gram test meal
- 5 grams of chia seeds (Experimental): 3 cookies (30 grams)
  Interventions: Other: 140 calories per 30 gram test meal
- 7 grams of chia seeds (Experimental): 3 cookies (30 grams)
  Interventions: Other: 140 calories per 30 gram test meal

INTERVENTIONS:
Other: 140 calories per 30 gram test meal — Food

SUMMARY:
To compare subjective appetite, satiety and glycemic responses for 3 h after consumption of investigational products containing 0, 3, 5 and 7 grams of chia seeds, controlling for energy intake. The primary objective is to compare total area under the curves (tAUC) of hunger and fullness ratings. The hypothesis is that chia seeds have a significant effect on hunger and/or fullness.

DETAILED DESCRIPTION:
Current nutrition guidelines in the United States and Canada recommend meeting protein needs with nutrient-dense foods among which include legumes, nuts, and seeds. Chia seeds are very high in dietary fiber, low in available-carbohydrate (avCHO), and good sources of alpha-linoleic acid, protein, and micronutrients. Chia has attracted interest as a functional food with studies showing several potential beneficial effects on health, among them their ability to increase satiety and/or reduce food intake. The effect on satiety of doses of chia less than 7g is not known. The primary objective of this study is to compare total area under the curves (tAUC) of hunger and fullness ratings for 3h after consumption among test-meals containing 0, 3, 5 and 7g of chia seeds, controlling for energy intake.

Secondary objectives are tAUC of desire to eat and prospective consumption, tAUC of average appetite, tAUC of subjective appetite ratings from 0-2, 2-3 and 0-3h, Effects of time and dose and the time×dose interaction of plasma glucose concentrations and increments for 3h after consuming the test products, Incremental area under the curve (iAUC) of plasma glucose over 0-2h, 2-3h and 0-3h, and Plasma glucose peak rise.

Main effects of chia dose, time, and the dose×time interaction will be examined. After demonstrating a significant interaction, individual endpoints will be assessed for the main effect of dose. The significance of differences between doses will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating, healthy individuals; at least n=45 aged 18-55 years and up to n=5 aged 56-65 years, inclusive
* BMI 18.5 to 34.9 kg/m², inclusive
* No history of diabetes mellitus
* Systolic blood pressure <160 mmHg and diastolic blood pressure <100 mmHg
* No major illness, trauma or surgery requiring hospitalization within 3 months of the screening visit
* Ability to understand the study procedures and willing to provide informed consent to participate in the study
* Subjects must be eligible to receive income in Canada and be covered by a health insurance plan such as OHIP
* Subjects are willing to follow current Covid guidelines with respect to attending study visits
* Subjects are willing to sign the informed consent prior to any procedures conducted

Exclusion Criteria:

* Participation in another PepsiCo trial in past 6 months
* Failure to meet any one of the inclusion criteria
* High alcohol consumption (>14 drinks per week and >4 drinks per day for males; and >7 drinks per week and >3 drinks per day for females), or history of alcohol or drug abuse.
* Individuals with a history of bariatric surgery, gastrointestinal disease, moderate or severe renal failure, moderate or severe liver disease or any other medical conditions or use of supplements or medications that increase risk to the subject or others or may affect the results, as judged by the Principal Investigator
* Unwillingness or inability to comply with the experimental procedures and to follow INQUIS safety guidelines
* Known intolerance, sensitivity, or allergy to any ingredients in the study test products.
* Subject is currently participating or recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement, or lifestyle modification.
* Reported weight change of > 5kg in the preceding 3 months
* History of an eating disorder (e.g., anorexia, bulimia, binge eating, pica, rumination, avoidant/restrictive food intake disorder)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Total area under the curve (tAUC) of hunger ratings among test-meals containing 0, 3, 5 and 7 grams of chia seeds. | Change from Time 0 -5 min (fasted) to +15, 30, 45, 60, 90, 120, 150 and 180 minutes after starting to eat
  Visual Analog Scale (VAS) Motivation to Eat Questionnaire, vertical mark on 100 mm line from 0=Not very hungry at all to 100= As hungry as I have ever felt
Total area under the curve (tAUC) of fullness ratings among test-meals containing 0, 3, 5 and 7 grams of chia seeds. | Change from Time 0 -5 min(fasted) to +15, 30, 45, 60, 90, 120, 150 and 180 minutes after starting to eat
  Visual Analog Scale (VAS) Motivation to Eat Questionnaire, vertical mark on 100 mm line from 0=Not full at all to 100=As full as I have ever felt

SECONDARY OUTCOMES:
Total area under the curve (tAUC) of desire to eat | Change from Time 0 -5 min (fasted) to +15, 30, 45, 60, 90, 120, 150 and 180 minutes after starting to eat
  Visual Analog Scale (VAS) Motivation to Eat Questionnaire, vertical mark on 100 mm line from 0=Very weak to 100=Very strong
Total area under the curve (tAUC) of prospective consumption | Change from Time 0 -5 min (fasted) to +15, 30, 45, 60, 90, 120, 150 and 180 minutes after starting to eat
  Visual Analog Scale (VAS) Motivation to Eat Questionnaire, vertical mark on100 mm line from 0=Nothing at all to 100= A large amount
Total area under the curve (tAUC) of average appetite | Change from Time 0 -5 minutes (fasted) to 2, 2-3 and 0-3 hours
  Average Appetite will be calculated as (Desire to Eat + Hunger + (100-Fullness) + Prospective consumption)/4
Total area under the curve (tAUC) of subjective appetite ratings | Change from Time 0 -5 minutes (fasted) to 2, 2-3 and 0-3 hours
  Measured using the Motivation to eat Visual Analog Scale (VAS) which consists of 4 questions assessing Desire to Eat, Hunger, Fullness, and Prospective Consumption
Effects of time and dose and the time × dose interaction of plasma glucose concentrations and increments | Change from Time 0 -5 min (fasted) to +15, 30, 45, 60, 90, 120, 150 and 180 minutes after starting to eat
  Main effects assessed using ANOVA. Differences between doses assessed using Tukey's test to adjust for multiple comparisons.
Incremental area under the curve (iAUC) of plasma glucose | Time 0 - 5 min (fasted) to 2, 2-3 and 0-3 hours after starting to eat
  Capillary blood via finger sticks centrifuged. Plasma glucose analyzed using a Vitros 350 Chemistry System
Plasma glucose peak rise | Time 0 -5 min (fasted) to +15, 30, 45, 60, 90, 120, 150 and 180 minutes after starting to eat
  The maximum glucose value

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No